CLINICAL TRIAL: NCT04839276
Title: The Effect of Administering Platelet-rich Fibrin to Autologous Fat Tissue in Injection Laryngoplasty for Unilateral Adductor Vocal Cord Paralysis
Brief Title: Administration of Platelet-rich Fibrin to Autologous Fat Tissue in Injection Laryngoplasty for Vocal Cord Paralysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: THT02
Record Dates: First submitted 2021-03-29; First posted 2021-04-09 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Vocal Cord Paralysis
Keywords: platelet-rich fibrin; vocal cord paralysis; dysphonia; injection laryngoplasty
MeSH Terms: conditions — Vocal Cord Paralysis; Dysphonia

STUDY DESIGN:
Intervention Model Description: The intervention group will receive injection laryngoplasty with a combination of PRF and microlobular autograph fat, while the control group will receive injection laryngoplasty with microlobular autograph fat.
Who Masked: Participant
Masking Description: The participants of the study know that they are being assigned to injection laryngoplasty procedures, but they didn't know whether PRF is being added to the autologous fat injection filler. The researchers are fully aware which participants are assigned to which procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injection Laryngoplasty with PRF and Autologous Fat (Experimental): Autologous microlobular fat is harvested from abdominal fat (area under the umbilical). 4 mL of microlobular fat is added to 4 mL of PRF and is smoothed by pushing it back and forth 15 times on a 2-tube 10 mL piston tube connected to a three-way connector. 3 mL of the mixture of fat and PRF is injected using a 12 G laryngoplasty syringe until medialization is achieved.
  Interventions: Combination Product: Injection Laryngoplasty with Platelet-rich Fibrin and Autologous Fat
- Injection Laryngoplasty with Autologous Fat (Active Comparator): Autologous microlobular fat is harvested from abdominal fat (area under the umbilical). 4 mL of microlobular fat is mashed by pushing it back and forth 15 times in a container of 2 piston tubes (10 mL) connected to a three-way connector. The crushed fat is injected as much as 3 mL using a 12 G laryngoplasty syringe until medialization is achieved.
  Interventions: Procedure: Injection Laryngoplasty with Autologous Fat

INTERVENTIONS:
Combination Product: Injection Laryngoplasty with Platelet-rich Fibrin and Autologous Fat — Injection Laryngoplasty with a combination of Platelet-rich Fibrin (PRF) and Autologous Fat. The PRF was made by taking 10 mL of peripheral blood from a healthy donor. Blood is then put inside the tube from the Regen lab kit. The tube was centrifuged with a force of 1,500 g (3000 rpm) for 5 minutes producing platelet-rich plasma (PRP). 4 mL of the aforementioned PRP was transferred to a 10 mL test tube, 1 M CaCl2 was added with a micropipette until final concentration of 25 mM was, reached producing PRF. Autologous fat harvested from the patient's abdomen was then mixed with the PRF solution to create the filler for injection laryngoplasty procedures. The injection procedures are done by placing the patient in a sniffing position followed by intraoral Kleinsasser laryngoscope insertion through the uvula, posterior pharyngeal wall, and epiglottis until the vocal cords are visible. Injection of the filler is then done to the paralyzed vocal cords.
  Other Names: RegenKit PRP Tube (Regen Lab)
  Arms: Injection Laryngoplasty with PRF and Autologous Fat
Procedure: Injection Laryngoplasty with Autologous Fat — Injection Laryngoplasty with autologous microlobular fat harvested from the patient's abdominal fat. Lidocaine was infiltrated under the umbilicus and then an incision was made in the area followed by fat removal using scissors. The fat was cleaned with 0.9% NaCl solution and then sheared into microlobular form. The injection procedures are done by placing the patient in a sniffing position followed by intraoral Kleinsasser laryngoscope insertion through the uvula, posterior pharyngeal wall, and epiglottis until the vocal cords are visible. Injection of the filler is then done to the paralyzed vocal cords.
  Other Names: Lipid Autograft
  Arms: Injection Laryngoplasty with Autologous Fat

SUMMARY:
The study tries to see the effect of using a combination of platelet-rich fibrin (PRF) and autologous fat as a filler for injection laryngoplasty procedures to treat unilateral adductor vocal cord paralysis.

DETAILED DESCRIPTION:
The vocal cord in humans is essential in producing voice used in communication and interaction between us. Vocal cord paralysis causes dysphonia, which interferes with communication, causing disruptions towards social activity and daily activities. One of the managements for vocal cord paralysis is medialisation and augmentation of the vocal cord through injection laryngoplasty. Autologous fat is one of the best fillers that can be used in this procedure, but it is highly absorbable and can be reabsorbed very quickly when injected to body tissues. Platelet Rich Fibrin (PRF) is a biomaterial consisting of growth factors that are thought to improve fat tissue longevity through increase of adipogenesis and angiogenesis. Improvement in fat longevity will improve clinical outcomes after laryngoplasty procedure potentially reducing number of repeated injections needed to achieve satisfactory resolution to vocal cord paralysis. The study evaluates a combination of PRF and autologous microlobular fat compared with autologous microlobular fat alone on laryngoplasty. Subjective evaluation was done by using Voice Handicap Index (VHI-30) questionnaire, while objective evaluation was conducted via computerized acoustic analysis/Multidimensional Voice Program (MDVP), videostroboscopy, and maximum phonation time.

ELIGIBILITY:
Inclusion Criteria:

* Subject is diagnosed with unilateral vocal cord paralysis in paramedian position or 3 months lateral onset without movement and mucosal waves of the vocal cords on videostroboscopy.
* Willing to give consent

Exclusion Criteria:

* Has a history of malignancy of the larynx or lung
* Subject isn't able to undergo injection laryngoplasty procedure under general anesthesia
* Subject with thrombositopenia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Voice Handicap Index-30 (VHI-30) questionnaire score | Before injection, 1 week, 4 week, 8 week post-injection
  The Voice Handicap Index Questionnaire-30 (VHI-30) is a subjective examination that can be used to assess the severity of voice disorders and their impact on social life. The VHI-30 categorizes handicaps into mild, moderate, and severe. This study assessed the VHI-30 score as a numerical scale so that the median value for the treatment and control groups can be obtained. The assessment was carried out based on the patient's perception by addressing complaints for each question (0 = never, 1 = almost never, 2 = sometimes, 3 = almost always, 4 = always). Patients with severe voice disorders will achieve a higher VHI-30 score. Interpretation of the total value of the VHI-30 includes mild disability values of 0 - 30; moderate disability of 31 - 60; and a severe disability of 61-120. Changes in VHI-30 score are recorded and statistically analysed.
Changes in Maximum Phonation Time | Before injection, 1 week, 4 week, 8 week post-injection
  Maximum phonation time describes the quality of the strength of the vocal cords when oscillating. The calculation of the phonation time will represent objective assessment of voice. Changes in maximum phonation time are recorded and statistically analysed.
Changes in Average Fundamental Frequency (F0) | Before injection, 1 week, 4 week, 8 week post-injection
  The Average Fundamental Frequency (F0) is a parameter in MDVP that represents the number of vocal cord vibration cycles in one second. The mean frequency ranges from 120 Hz for men and 200 Hz for women, but this is also influenced by age, smoking and accent language. The average fundamental frequency reflects the biochemical characteristics of the vocal cords when interacting with the air flow in its path, these biochemical properties are influenced by the structure of the larynx and muscle tone. Changes in F0 are recorded and statistically analysed.
Changes in Jitter and Shimmer | Before injection, 1 week, 4 week, 8 week post-injection
  Jitter and Shimmer is a parameter in MDVP that represents variations that occur in the basic frequency. Jitter denotes the chaos of sound wave frequency caused by a lack of control over the vibration of the vocal cords. Shimmer shows the chaos of sound wave amplitude which is influenced by decreased resistance of the glottis and presence of mass lesions of the vocal cords, associated with inadequate adduction of the vocal cords and irregularity of the surface of the vocal cords. Presence of jitter and shimmer denotes that there are disruption in phonation quality caused by problems in vocal cords. Changes in jitter and shimmer are recorded and statistically analysed.
Changes in Noise to Harmonic Ratio (NHR) | Before injection, 1 week, 4 week, 8 week post-injection
  NHR is a parameter in MDVP that represents ratio of non-harmonic and harmonic waves in a certain sound wave period. NHR describes the quality of the amount of noise in the sound. Inadequate closure of the vocal cords and periodic vibrations of the vocal cords cause excessive air flow as it passes through the vocal cords, causing turbulence and noise. Normal and periodic sound signals will have a small NHR, while dysphonia sound signals will have a large NHR value. Changes in NHR are recorded and statistically analysed.
Changes in Voice Turbulence Index (VTI) | Before injection, 1 week, 4 week, 8 week post-injection
  VTI (Voice Turbulence Index) is a parameter in MDVP that represents the ratio between non-harmonic waves at high frequencies of 2800 - 5800 Hz and harmonic waves at frequencies of 70 - 4500 Hz. This parameter assesses the energy level of high frequency noise and is largely related to the turbulence of sound caused due to loss of adduction motion. This parameter also relates to variations in the frequency or amplitude of sound, where the turbulence of sound occurs due to changes in muscle control. Changes in VTI are recorded and statistically analysed.
Changes in Amplitude Tremor Intensity Index (ATRI) | Before injection, 1 week, 4 week, 8 week post-injection
  ATRI is a parameter in MDVP that represents the mean ratio of the low frequency amplitude to the total amplitude of the sound being examined. This parameter indicates the stability and strength of the vocal cords during phonation. Changes in ATRI are recorded and statistically analysed.
Changes in Vocal Cord Closure Pattern | Before injection, 1 week, 4 week, 8 week post-injection
  The closure pattern of the vocal cords is one of the parameters in videostroboscopy. This examination looks at the pattern and medial edge of the vocal cords when closed and insulated. Changes in Vocal Cord Closure Pattern are recorded and statistically analysed.
Changes in Amplitude | Before injection, 1 week, 4 week, 8 week post-injection
  The amplitude is one of the parameters in videostroboscopy. Amplitude is the amount of horizontal movement of the vocal cords. The magnitude of the amplitude is assessed by dividing the horizontal line into 5 sections from medial to lateral of the vocal cords. Changes in amplitude are recorded and statistically analysed.
Changes in Mucosal Waves | Before injection, 1 week, 4 week, 8 week post-injection
  The mucosal waves is one of the parameters in videostroboscopy. Mucosal waves are the movement of the vocal cords from an inferior to a superior direction following the glottic cycle on the vertical axis. Changes in mucosal waves are recorded and statistically analysed.
Changes in Vertical Level | Before injection, 1 week, 4 week, 8 week post-injection
  The vertical level is a parameter of the vocal cords on videostroboscopy that describes the difference in the height of the vocal cords that meet and are seen in the medial of the vocal cords. Changes in vertical level are recorded and statistically analysed.
Changes in Supraglottic Activity | Before injection, 1 week, 4 week, 8 week post-injection
  The supraglottic activity is one of the parameters in videostroboscopy. Supraglottic activity describes a narrowing of the supraglottic structure wherein one of them is a collapsed arytenoid. Changes in supraglottic activity are recorded and statistically analysed.
Changes in Non-vibrating Parts | Before injection, 1 week, 4 week, 8 week post-injection
  The non-vibrating parts is one of the parameters in videostroboscopy. The non-vibrating part is the part of the vocal cords that does not experience vibrations due to tissue rigidity. Assessment of this parameter is by dividing the right and left vocal cords into 10 regions each with an oval line. Changes in non-vibrating parts are recorded and statistically analysed.
Changes in Free Edge Contours | Before injection, 1 week, 4 week, 8 week post-injection
  The free edge contours is one of the parameters in videostroboscopy. This parameter represents the free edge of the medial side of the vocal cords at maximal abduction. Changes in free edge contours are recorded and statistically analysed.
Changes in Symmetrical Pattern | Before injection, 1 week, 4 week, 8 week post-injection
  This parameter assesses the symmetrical movement of the right and left vocal cords during oscillation using videostroboscopy. The results of the assessment on this parameter are symmetrical or asymmetrical. Changes in symmetrical pattern are recorded and statistically analysed.
Changes in Closure Phase | Before injection, 1 week, 4 week, 8 week post-injection
  The closure phase is a parameter that compares the amount of closure and opening of the vocal cords in one glottic cycle. Assessment is done by looking at a collection of pictures from videostroboscopy when the vocal cords oscillate. Changes in closure phase are recorded and statistically analysed.
Changes in The Stability of The Vocal Cords | Before injection, 1 week, 4 week, 8 week post-injection
  The stability of the vocal cords is a parameter that measures the vibration and amplitude of the vocal cords that are oscillating in one glottic cycle Assessment of this parameter where done through videostroboscopy. Changes in the stability of the vocal cords are recorded and statistically analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Mirta H Reksodiputro, SpTHT-KL(K), Study Chair — Department of ENT, Faculty of Medicine, University of Indonesia; Syahrial M Hutauruk, SpTHT-KL(K), Study Chair — Department of ENT, Faculty of Medicine, University of Indonesia; Trimartani Koento, SpTHT-KL(K), Study Chair — Department of ENT, Faculty of Medicine, University of Indonesia; Fauziah Fardizza, SpTHT-KL(K), Study Chair — Department of ENT, Faculty of Medicine, University of Indonesia; Razki YM Hakim, SpTHT-KL, Principal Investigator — Department of ENT, Faculty of Medicine, University of Indonesia; Sacha Audindra, M.D, BMedSci, Principal Investigator — Department of ENT, Faculty of Medicine, University of Indonesia; Mikhael Yosia, M.D, DTM&H, Principal Investigator — Department of ENT, Faculty of Medicine, University of Indonesia
Locations (1):
- Fakultas Kedokteran Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stachler RJ, Francis DO, Schwartz SR, Damask CC, Digoy GP, Krouse HJ, McCoy SJ, Ouellette DR, Patel RR, Reavis CCW, Smith LJ, Smith M, Strode SW, Woo P, Nnacheta LC. Clinical Practice Guideline: Hoarseness (Dysphonia) (Update) Executive Summary. Otolaryngol Head Neck Surg. 2018 Mar;158(3):409-426. doi: 10.1177/0194599817751031. PMID 29494316
- [Background] Rubin AD, Sataloff RT. Vocal fold paresis and paralysis. Otolaryngol Clin North Am. 2007 Oct;40(5):1109-31, viii-ix. doi: 10.1016/j.otc.2007.05.012. PMID 17765698
- [Background] Mattei A, Desuter G, Roux M, Lee BJ, Louges MA, Osipenko E, Sadoughi B, Schneider-Stickler B, Fanous A, Giovanni A. International consensus (ICON) on basic voice assessment for unilateral vocal fold paralysis. Eur Ann Otorhinolaryngol Head Neck Dis. 2018 Feb;135(1S):S11-S15. doi: 10.1016/j.anorl.2017.12.007. Epub 2018 Feb 3. PMID 29398504
- [Background] Seyed Toutounchi SJ, Eydi M, Golzari SE, Ghaffari MR, Parvizian N. Vocal cord paralysis and its etiologies: a prospective study. J Cardiovasc Thorac Res. 2014;6(1):47-50. doi: 10.5681/jcvtr.2014.009. Epub 2014 Mar 4. PMID 24753832
- [Background] Kwon TK, Buckmire R. Injection laryngoplasty for management of unilateral vocal fold paralysis. Curr Opin Otolaryngol Head Neck Surg. 2004 Dec;12(6):538-42. doi: 10.1097/01.moo.0000144393.40874.98. PMID 15548914
- [Background] Graboyes EM, Bradley JP, Meyers BF, Nussenbaum B. Efficacy and safety of acute injection laryngoplasty for vocal cord paralysis following thoracic surgery. Laryngoscope. 2011 Nov;121(11):2406-10. doi: 10.1002/lary.22178. Epub 2011 Oct 12. PMID 21994176